CLINICAL TRIAL: NCT05261971
Title: Evaluation of the Effects of Treatments Applied to Patients With Facial Myalgia on Quality of Life and Occlusion Parameters
Brief Title: Evaluation of the Effects of Treatments Applied to Patients With Facial Myalgia on Occlusion Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Beyza Ünalan Değirmenci, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21.11.2018/01
Record Dates: First submitted 2022-02-17; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Occlusion; Quality of Life
Keywords: T Scan; Facial Myalgia
MeSH Terms: conditions — Bites and Stings | interventions — Etodolac; thiocolchicoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medical therapy (No Intervention): One non-steroidal anti-inflammatory drug (400mg etodolac) and one muscle relaxant drug (4 mg thiocolchicoside) were prescribed to the patients in this group.
- Hard Splint Therapy (Active Comparator): The patients in this group were asked to use a hard splint delivered to them to use at night.
  Interventions: Drug: Etodolac 400 MG; Drug: Thiocolchicoside
- Soft Splint Therapy (Active Comparator): The patients in this group were asked to use a soft splint delivered to them to use at night.
  Interventions: Drug: Etodolac 400 MG; Drug: Thiocolchicoside

INTERVENTIONS:
Drug: Etodolac 400 MG — Patients were asked to drink a tablet containing 400 mg of etodolac every 24 hours with a glass of water.
  Other Names: Etol Fort
  Arms: Hard Splint Therapy; Soft Splint Therapy
Drug: Thiocolchicoside — Patients were asked to drink a tablet containing 4 mg of thiocolchicoside every 24 hours with a glass of water.
  Other Names: Muscoflex
  Arms: Hard Splint Therapy; Soft Splint Therapy

SUMMARY:
The temporomandibular joint (TMJ) is closely related to neuromuscular components. A problem occurring in any of these components or parts of the TMJ interferes with the harmonic functioning of the TMJ and invites temporomandibular joint disorders (TMD).Management of TMD can be conservative or surgical. Physiotherapy, local steam application, external muscle massage, occlusal adjustment, analgesic and physiotherapeutic medication and splint treatments are the most frequently recommended conservative treatments. Today, occlusal adjustments are made with the help of a prosthetic or orthodontic appliance. With these intraorally used occlusal splints, a balanced occlusal contact is achieved without applying any force to the mandible in the resting position. Occlusal splints are available in different designs and different construction materials. The stabilization splint, which is one of the most frequently used occlusal splints, and the modified Hawley splint are appliances produced from hard materials. However, some researchers have commented that soft splints produced from resilient materials may also be useful in the distribution of excessive force formed in parafunctional habits. While there are studies stating that hard splints provide more successful results than soft splints in functional problems of the chewing system, there are also studies reporting that they have similar efficacy on muscle pain after short-term use. However, there are no studies in the literature that compare their efficacy in short-term and long-term myalgia patients and demonstrate their efficacy using an objective test such as digital occlusion analysis. There was no study on the effectiveness of different splints on the patient's quality of life. It would be appropriate to carry out our study to fill this gap in the literature.The main purpose of this study is to digitally examine and compare the effects of three different treatment methods (medical therapy, medical therapy+soft splint, medical therapy +hard splint) applied to patients diagnosed with facial myalgia after temporomandibular joint examination on the existing occlusion changes.

ELIGIBILITY:
Inclusion Criteria:

* No systemic disease that may have effects on masticatory muscles or TMJ
* Individuals who do not have any tooth loss other than molar teeth and accept the treatments to be performed.

Exclusion Criteria:

* Individuals with total or partial prosthesis with distal extension
* Individuals who have previously received medical, pharmacological or any type of treatment for TMD
* Individuals who have recently been exposed to facial or cervical trauma
* Individuals with the syndrome who have the potential to affect any component of the stomatognathic system
* Individuals with parafunctional habits such as clenching or grinding their teeth.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-04-12 (Actual)

PRIMARY OUTCOMES:
Effects of treatment method on occlusion time parameters | 1 week- 6 month
  Occlusion times, left and right lateral disclusion times and protrusive disclusion times are among the occlusion parameters. In each control session, researchers will record these parameters in seconds using the T-Scan III system.
Effects of treatment method on distribution of right-left occlusion force percentages | 1 week- 6 month
  In each control session, researchers will record these parameters as percentages using the T-Scan III system.

CONTACTS AND LOCATIONS:
Locations (1):
- Beyza Ünalan Değirmenci, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If requested from the principal investigator, information will be shared via e-mail without time limit.
Supporting Information: Study Protocol
Time Frame: If requested from the principal investigator, information will be shared via e-mail without time limit.
Access Criteria: If requested from the principal investigator, information will be shared via e-mail without time limit.

REFERENCES:
- [Background] Dworkin SF, Huggins KH, Wilson L, Mancl L, Turner J, Massoth D, LeResche L, Truelove E. A randomized clinical trial using research diagnostic criteria for temporomandibular disorders-axis II to target clinic cases for a tailored self-care TMD treatment program. J Orofac Pain. 2002 Winter;16(1):48-63. PMID 11889659
- [Background] Dworkin SF, LeResche L. Research diagnostic criteria for temporomandibular disorders: review, criteria, examinations and specifications, critique. J Craniomandib Disord. 1992 Fall;6(4):301-55. No abstract available. PMID 1298767
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Seifeldin SA, Elhayes KA. Soft versus hard occlusal splint therapy in the management of temporomandibular disorders (TMDs). Saudi Dent J. 2015 Oct;27(4):208-14. doi: 10.1016/j.sdentj.2014.12.004. Epub 2015 Jun 25. PMID 26644756
- [Background] Nagata K, Maruyama H, Mizuhashi R, Morita S, Hori S, Yokoe T, Sugawara Y. Efficacy of stabilisation splint therapy combined with non-splint multimodal therapy for treating RDC/TMD axis I patients: a randomised controlled trial. J Oral Rehabil. 2015 Dec;42(12):890-9. doi: 10.1111/joor.12332. Epub 2015 Jul 14. PMID 26174571